CLINICAL TRIAL: NCT06285734
Title: Clinical Characteristics of Small Intestinal Bacterial Overgrowth in Individuals with Abdominal Distention
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Qilu Hospital of Shandong University (Qingdao) (Other); Jinan Central Hospital (Other); Zaozhuang Municipal Hospital (Other); Weihai Municipal Hospital (Other); Central Hospital of Zibo (Other); Weifang People's Hospital (Other); Dezhou Hospital Qilu Hospital of Shandong University (Other); Binzhou Medical University (Other); Qihe Xian Renmin Hospital (Unknown)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital, Shandong University
Other Study IDs: KYLL-202312-049
Record Dates: First submitted 2024-02-05; First posted 2024-02-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Distention
Keywords: abdominal distention; small intestinal bacterial overgrowth; orocecal transit time; cross-sectional survey
MeSH Terms: interventions — Breath Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The exhaled air of the patient after taking the substrate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Breath test — The concentration of methane and hydrogen in the exhaled gas of patients with Abdominal distention is measured by a breath test to determine the presence of SIBO and abnormal OCTT.

SUMMARY:
Abdominal distention represents a prevalent clinical manifestation characterized by an unclear etiology and pathogenesis. This symptomatology is frequently observed in various conditions, including small intestinal bacterial overgrowth (SIBO) and abnormal orocecal transit time (OCTT). The utilization of the breath test as a non-invasive diagnostic approach has become widespread in recent years for identifying SIBO and abnormalities in OCTT. In this study, the prevalence of SIBO and OCTT irregularities in individuals presenting with abdominal distention was ascertained through the implementation of the breath test. Furthermore, the correlation between abdominal distention and SIBO/OCTT was analysed to enhance the elucidation of the underlying etiology of abdominal distention. These findings aim to offer valuable insights for refining clinical comprehension and strategies related to the diagnosis and treatment of abdominal distention.

DETAILED DESCRIPTION:
Abdominal distention represents a prevalent clinical manifestation characterized by an unclear etiology and pathogenesis. And the prevalence of abdominal distension is high in the population. This symptomatology is frequently observed in various conditions, including small intestinal bacterial overgrowth (SIBO) and abnormal orocecal transit time (OCTT). The utilization of the breath test as a non-invasive diagnostic approach has become widespread in recent years for identifying SIBO and abnormalities in OCTT. In this study, the prevalence of SIBO and OCTT irregularities in individuals presenting with abdominal distention was ascertained through the implementation of the breath test. Furthermore, the correlation between the clinical features such as severity, location, and frequency of abdominal distension and SIBO/OCTT was analysed to enhance the elucidation of the underlying etiology of abdominal distention. These findings aim to offer valuable insights for refining clinical comprehension and strategies related to the diagnosis and treatment of abdominal distention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70 years.
2. Patients presenting with the primary complaint of abdominal bloating and/or abdominal distension, or those exhibiting abdominal distension with prominence over other symptoms.

Exclusion Criteria:

1. Patients who are pregnant or lactating.
2. Patients have history of gastrointestinal malignancy or gastrointestinal surgery.
3. Patients manifesting food intolerance or presenting with a confirmed diagnosis or suspicion of lactose intolerance.
4. Patients with urinary system (chronic kidney disease, etc.), immune system (scleroderma, etc.), nervous system (Parkinson's disease, etc.), mental system (depression, etc.), or other diseases outside the digestive system.
5. Patients who used antibiotics or microecological agents or underwent endoscopic examination within two weeks.
6. Patients with a medication history encompassing motility enhancers, secretory enhancers, antifoaming agents, spasmolytics, opioids, and antidepressants within the past week.
7. Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Abdominal distension patients in the outpatient department at Qilu Hospital of Shandong University.
Sampling Method: Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Positive rate of SIBO in patients with abdominal distension | 2024-03-01 to 2025-08-01
  Detect the positive rate of SIBO in patients with abdominal distension by breath test

SECONDARY OUTCOMES:
Positive rate of abnormal OCTT in patients with abdominal distension | 2024-03-01 to 2025-08-01
  Detect the positive rate of abnormal OCTT in patients with abdominal distension by breath test
Correlation between clinical features of patients with abdominal distension and SIBO | 2024-03-01 to 2025-08-01
  Analyze the correlation between clinical features of patients with abdominal distension and SIBO
Correlation between clinical features of patients with abdominal distension and OCTT | 2024-03-01 to 2025-08-01
  Analyze the correlation between clinical features of patients with abdominal distension and OCTT

CONTACTS AND LOCATIONS:
Overall Officials: Feixue Chen, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Gastroenterology Department of Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No